CLINICAL TRIAL: NCT02297685
Title: Effectiveness of Two Electrotherapy Techniques to Treat Chronic Low Back Pain
Brief Title: Effectiveness of Electrotherapy Techniques to Treat Low Back Pain
Acronym: TENBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Collaborators: Public Health Service of Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCJC-15
Record Dates: First submitted 2014-11-17; First posted 2014-11-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Chronic Low Back Pain
Keywords: Transcutaneous electrical nerve stimulation (TENS); Interferential currents therapy; Therapeutic exercises; Low back pain; Rehabilitation
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham Transcutaneous nerve stimulation (Sham Comparator): The group with sham TENS did not receive any current. Four surface electrodes (5×5 cm Prim-Trode®, Spain) were symmetrically placed over the L1 and L5 transverse processes with respect to the spine. The patients were informed that they may or may not feel any sensation at the application site of the electrodes.
  Interventions: Device: Sham Transcutaneous nerve stimulation
- Transcutaneous nerve stimulation (Experimental): The group with TENS received current at a frequency of 80 Hz and with a pulse width of 150 μs with two channels, for 30 minutes over a period of 4 weeks, including a total of 12 sessions.
  Interventions: Device: Transcutaneous nerve stimulation
- Interferential currents (Experimental): The group with IC received a base frequency of 4000 Hz with AMF = 65 Hz, sweep = 95 Hz and slope of 1/1 in tetrapolar mode, for 30 minutes over a period of 4 weeks, including a total of 12 sessions.
  Interventions: Device: Interferential currents

INTERVENTIONS:
Device: Sham Transcutaneous nerve stimulation — The group with sham transcutaneous nerve stimulation (TENS) did not receive any electrical treatment. We placed 4 surface electrodes (5x5 cm Prim-Trode, Spain) over the L1 and L5 transverse processes with respect to the spine but we did not delivery any current. The patients were informed that they may or may not feel any sensation at the application site of the electrodes.
  Other Names: Sham TENS
  Arms: Sham Transcutaneous nerve stimulation
Device: Transcutaneous nerve stimulation — The group with transcutaneous nerve stimulation (TENS) received electrical stimulation for 12 sessions at a frequency of 80 Hz and with a pulse width of 150 ns. The TENS was delivered by using 4 surface electrodes (5x5 cm Prim-Trode, Spain) placed over the L1 and L5 transverse processes with respect to the spine. The current intensity was set 3 times during each session according to each patient's sensitivity.
  Other Names: TENS
  Arms: Transcutaneous nerve stimulation
Device: Interferential currents — The group with IC received a base frequency of 4000 Hz with AMF = 65 Hz, sweep = 95 Hz and slope of 1/1 in tetrapolar mode (Endomed 492 Enraf-nonius, Netherlands). The current was applied by using 4 surface electrodes (5x5 cm Prim-Trode, Spain) into two channels: were symmetrically placed over the L1 and L5 transverse processes with respect to the spine; the current intensity was set 3 times during each session according to each patient's sensitivity.
  Other Names: IC
  Arms: Interferential currents

SUMMARY:
Objective: The aim of this investigation was compare the effectiveness of transcutaneous electrical nerve stimulation (TENS) and interferential currents (IC) on chronic low back pain. Forty-eight patients diagnosed as having chronic low back pain were randomly assigned to three groups: control (sham electrotherapy; age 47 ± 8 years), interferential currents (IC; age 48 ± 8 years) and transcutaneous electrical nerve stimulation (TENS; age 48 ± 8 years). Patients in all groups received 12 × 30-min sessions of the assigned treatment for a period of 4 weeks plus therapeutic exercises. Before and after the treatment, low back pain was measured using a 100-mm visual analogue scale and functional disability level was measured using the Rolland Morris Disability Questionnaire. Participants status was followed up 3 months after the end of the treatment.

DETAILED DESCRIPTION:
Subjects

The subjects for this study were recruited from a waiting list at the Almendrales Physiotherapy Center (Madrid, Spain). Potential participants had to be older than 18 years and present continuous low back pain for more than 12 weeks. Potential participants were then examined by an independent specialist and the diagnosis of LBP was made according the medical diagnosis, the Roland Morris Disability Questionnaire (RMQD)24 and an X-ray. With these inclusion criteria, a total of 96 patients were contacted to participate in the experiment. Twenty-one participants were excluded because they fulfilled one or several of the following exclusion criteria: individuals presenting trauma, disc disease or lumbosciaticas; individuals who were receiving pain-relieving treatments with another physiotherapy method at the same time; patients with previous surgery or intra-articular injections; individuals with contraindications against electrotherapy; and declined to participate.

Treatment groups

The experimental design was a randomized, double-blind sham-controlled clinical trial. After the preliminary examination, 48 patients were randomly assigned to three groups: control (sham electrotherapy), transcutaneous electrical nerve stimulation (TENS) and interferential currents (IC). A set of sealed and sequentially numbered opaque envelopes was used for group assignment. The study was double-blind because the examiner had no contact with the patient during the duration of the treatment and patients were not informed about the electrotherapy technique they received during the investigation.

Intervention

Each treatment was applied 3 times per week on alternate days (excluding weekends) over a period of 4 weeks, including a total of 12 sessions. All the treatments were administered by an experienced physiotherapist. Four surface electrodes (5×5 cm Prim-Trode®, Spain) were symmetrically placed over the L1 and L5 transverse processes with respect to the spine; the current intensity was set 3 times during each session according to each patient's sensitivity. The patients were informed that they may or may not feel any sensation at the application site of the electrodes. The group with IC received a base frequency of 4000 Hz with AMF = 65 Hz, sweep = 95 Hz and slope of 1/1 in tetrapolar mode (Endomed 492 Enraf-nonius, Netherlands). The group with TENS received current at a frequency of 80 Hz and with a pulse width of 150 μs with two channels (P-82 TENS med Enraf-nonius, Netherlands). Participants in the control group received the same procedures (e.g., electrode placement) but the current was always equal to 0. In each session, the electrical stimulation technique was administered for 30 minutes while the subjects were comfortable seated in an adjustable chair. After the electrostimulation procedures, all participants performed a 30-min session of therapeutic exercises. The session included lumbar stabilization (5 different exercises) and conventional stretching (5 different exercises). Each exercise was performed for 10 repetitions and with 60 s of rest between exercises. These exercise routines were added to the all the electrotherapy techniques investigated at the request of the Ethics Committee in order to provide treatment to all participants.

Outcome measurements

The day before the onset of the treatment (pre-treatment) and the day after the end of the treatment (post-treatment), the intensity of low back pain was evaluated by using a 100-mm visual analogue pain scale (VAS). The functional status of each individual was measured using the Rolland Morris Disability Questionnaire(RMDQ) at these same time-points. The RMDQ is a simple, fast and valid questionnaire to assess the LBP disability. It consists of 24 items that reflect limitation in different activities of daily living attributed by the patient to low back pain. Each item receives a score of 1 point, so the RMDQ score ranges between 0 (no disability) and 24 points (the maximum possible disability). The use of disability scales, such as RMDQ, has been shown to correlate with physical incapacity better than the scales that measure the intensity of pain, X Rays, magnetic resonance imaging scans (MRIs), and computerized tomography scans.

The straight leg raise (SLR) in both legs was also used to measure the range of motion of the leg. For this measurement, an inclinometer (Baseline, Enterprises Inc., USA) was applied to the anterior tibial tuberosity with the patient lying on a treatment stretcher. To prevent the external rotation of the hip, the contralateral leg was fixed with a strap to the stretcher. The examiner passively flexed the participant's hip with the knee fully extended until the subject felt tightness in the hamstring area or until the lower back was destabilized. The SLR (in degrees) was calculated separately for each leg by using one repetition.

Pressure pain threshold (PPT) was measured at the lumbosacral joint and at the right and left sacroiliac joints with the application of a pressure algometer (FPK 20, Wagner Instruments, USA) with a rubber tip of 1 cm2. The PPT recorded the maximal pressure (kg/cm2) applied until the participant perceived it as painful. The PPT measured at each location was repeated three times with 1 min of rest between repetitions. The average value of these 3 measurements was used for further analysis.

Three months after the end of the treatments, the RMDQ was applied to all participants to evaluate the LBP disability and the maintenance of the improvements obtained by the treatments. The follow-up was performed by the same independent experimenter and in the same experimental conditions.

Statistical analysis

All the data were analyzed using the SPSS v.20 statistical package. Descriptive statistics were calculated for each group (mean and standard deviation). Normality was tested with the Shapiro-Wilk test. All the variables presented a normal distribution in this test (P > 0.05). Baseline characteristics were compared using the analysis of variance (ANOVA) for measuring independent data. Pre-to-post treatment changes and the comparison between groups were performed by using a two-way ANOVA (group x time). After a significant F test, differences between means were identified using Tukey's HSD post hoc procedure. The level of significance was established at P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* The subjects for this study were recruited from a waiting list from patients with acute low back pain.
* To be included in the list they had to be older than 18 years and have had unilateral shoulder pain for more than 12 weeks.
* Potential participants were then examined by an independent specialist and the diagnosis of LBP was made according to the Roland Morris Disability Questionnaire."

Exclusion Criteria:

* The following participants were excluded from the investigation: individuals presenting trauma, disc disease or lumbosciaticas; individuals who were receiving pain-relieving treatments with another physiotherapy method at the same time; patients with previous surgery or intra-articular injections; individuals with contraindications against electrotherapy and those who declined to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
Functional status | Change after 3 weeks of electrotherpy treatment
  The functional status of each individual was measured using the Rolland Morris Disability Questionnaire (RMDQ) before and after 3 weeks of eletrotherapy treatment. The RMDQ is a simple, fast and valid questionnaire to assess the LBP disability. It consists of 24 items that reflect limitation in different activities of daily living attributed by the patient to low back pain. Each item receives a score of 1 point, so the RMDQ score ranges between 0 (no disability) and 24 points (the maximum possible disability)
Perceptual evaluation of low back pain | Change after 3 weeks of electrotherpy treatment
  The intensity of low back pain was evaluated before and after 3 weeks of electrotherpy treatment by using a 100-mm visual analogue pain scale (VAS)
The straight leg raise (SLR) | Change after 3 weeks of electrotherpy treatment
  The straight leg raise (SLR) in both legs was also used to measure the range of motion of the leg. For this measurement, an inclinometer (Baseline, Enterprises Inc., USA) was applied to the anterior tibial tuberosity with the patient lying on a treatment stretcher. To prevent the external rotation of the hip, the contralateral leg was fixed with a strap to the stretcher. The examiner passively flexed the participant's hip with the knee fully extended until the subject felt tightness in the hamstring area or until the lower back was destabilized. The SLR (in degrees) was calculated separately for each leg by using one repetition.
Pressure pain threshold (PPT) | Change after 3 weeks of electrotherpy treatment
  Pressure pain threshold (PPT) was measured at the lumbosacral joint and at the right and left sacroiliac joints with the application of a pressure algometer (FPK 20, Wagner Instruments, USA) with a rubber tip of 1 cm2. The PPT recorded the maximal pressure (kg/cm2) applied until the participant perceived it as painful. The PPT measured at each location was repeated three times with 1 min of rest between repetitions. The average value of these 3 measurements was used for further analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Del Coso, PhD, Principal Investigator — Camilo Jose Cela University
Locations (1):
- Health Center Almendrales, Madrid, Spain

REFERENCES:
- [Background] Thiese MS, Hughes M, Biggs J. Electrical stimulation for chronic non-specific low back pain in a working-age population: a 12-week double blinded randomized controlled trial. BMC Musculoskelet Disord. 2013 Mar 28;14:117. doi: 10.1186/1471-2474-14-117. PMID 23537462